CLINICAL TRIAL: NCT03640767
Title: The Effectiveness of Text Message-based Rehabilitation Program on Cardiometabolic Risk Factors for Patients With Peripheral Artery Disease Post-surgical Revascularization: A Randomized Controlled Trial
Brief Title: Effectiveness of Text Message-based Rehabilitation Program for Patients With Peripheral Artery Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Caritas Institute of Higher Education (Other)
Responsible Party: Principal Investigator, Choy Hau Kim, Senior Lecturer, Caritas Institute of Higher Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HRE170101
Record Dates: First submitted 2018-08-13; First posted 2018-08-21 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Message-based Rehabilitation for Peripheral Artery Disease Patients
Keywords: Rehabilitation; Peripheral artery disease; Mobile phone text message
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: This pilot randomised controlled trial aimed at examining the effectiveness of message-based lifestyle intervention. Peripheral artery disease patients who have received revascularization in the past 6 months, are randomized into 2 groups. The total sample size will be 160.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- message-based lifestyle intervention (Experimental): The intervention group will receive 4 mobile phone messages per week for 24 weeks.
  Interventions: Behavioral: Message-based lifestyle intervention
- Control (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Message-based lifestyle intervention — Peripheral artery disease patients who have received revascularization in the past 6 months, are randomized into 2 groups. The total sample size will be 160. Both intervention and control groups will receive face-to-face lifestyle adherence counseling and booklets at baseline. The intervention group will receive 4 mobile phone messages per week for 24 weeks. The messages are motivational advice to support lifestyle behavioral modification in various stages of behavioral changes.
  Arms: message-based lifestyle intervention

SUMMARY:
Background: Many patients with peripheral artery disease are unable to achieve healthy lifestyle after revascularization. There is evidence that rehabilitation program could result in decreased re-admission, reduced cardiometabolic risk factors and improved quality of life.

Aim: This first randomized controlled trial to examine the effectiveness of mobile phone text message-based rehabilitation on low density lipoprotein (LDL), Ankle Brachial Index (ABI), healthy lifestyle behaviors and quality of life for patients after revascularization. Methods: This is a 6 months randomized controlled trial. It is hypothesized that message-based rehabilitation program will be effective in improving the low density lipoprotein (LDL), Ankle Brachial Index (ABI), healthy lifestyle behaviors and quality of life for patients with peripheral artery disease after surgical revascularization. A total of 160 participants will be recruited for the study. The participants will be randomly divided into intervention and control groups. Both intervention and control groups will receive face-to-face lifestyle adherence counseling and booklet at baseline. The intervention group will receive 4 mobile phone messages per week for 24 weeks.

All participants will be asked to fill in the questionnaires at the baseline, 6-week and 6-month follow-up in Surgical Out Patient Department (SOPD). Participants' blood results of low density lipoprotein (LDL) at the baseline and at 6-month follow-up will be retrieved from Computer Management System in SOPD The primary outcomes are the fasting LDL levels at 6 months. Secondary outcome are Ankle-Brachial Index (ABI), BMI, Fasting glucose level, HDL level, Total cholesterol level, self-reported adherence to healthy lifestyle behaviours, quality of life and smoking status.

Participants: The target participants of this study are peripheral artery disease patients who have received revascularization in the Surgical Department of a regional hospital in Hong Kong. The eligible participants are Chinese, aged 50 years or above, and with medical record of peripheral artery disease with revascularization done in the past 6 months. The participants should be able to receive and read Chinese texts from their own mobile phones and are available to come back for a 6-month follow-up for lifestyle counselling. The potential participants will be excluded if they refuse to provide an informed-consent form or if they have medical records stating their lack of capacity to provide informed consent. The recruitment procedure will take place in Department of Surgery in a regional hospital.

Study setting: The study will be conducted in the Surgical Department of a regional hospital in Hong Kong.

DETAILED DESCRIPTION:
Background Peripheral artery disease (PAD) is a circulatory disease which associated with narrowing of arteries in the lower limbs. It is also a common atherosclerotic vascular disease affecting 3-12% of the global population [1]. With aging of the global population and increasing industrialization, PAD is expected to increase further in the next few decades. Worse of all, PAD increases risk of coronary, cerebrovascular complication including death [2]. So secondary prevention is essential for patients with PAD especially after revascularization.

There is robust evidence that the secondary prevention of peripheral artery disease can be achieved by lifestyle modification [3-4]. The American Heart Association (AHA) recommended that smoking cessation, glycemic control and structured exercise are import elements of care for patient with PAD [5]. Despite the need of secondary prevention and the evidence-based guidelines from AHA, there is no structured rehabilitation program for PAD patients in Hong Kong. Recent studies reported secondary prevention of PAD mainly focus on exercise and medication therapy. However, a single lifestyle behavioral change could not address the needs of the patients who have multiple lifestyle risk factors. Since many PAD patients have more than one lifestyle risk factor, the rehabilitation program targeting multiple lifestyle behavioral changes will be more benefit to the at risk patients.

Mobile-rehabilitation is a new concept to deliver the rehabilitation program. Center-based rehabilitation is well evidenced to reduce mortality, unplanned hospital admissions and improve quality of life and psychological well-being of the patients [6]. However, its benefits is limited by low referral rate and inaccessibility of program site [7]. Mobile phone messaging can be used to motivate and reinforce the lifestyle behavioral changes. It can also prevent patients from relapsing to the previous unhealthy lifestyle behavioral stage. Current studies show a positive result of using texting to promote healthy lifestyle behaviors among adults with cardiovascular disease [8-9]. Considering that the mobile-phone penetration rate in Hong Kong is about 96.1% [10], the use of texting can be an innovative and cost-effective tool to promote a healthy lifestyle and improve quality of life of PAD patients.

To the best of the author's knowledge, there have been no Randomized Controlled Trial (RCT) of a stand-alone mobile phone message-based rehabilitation program designed to help peripheral artery disease patients. This is the first randomized controlled trial to examine the effectiveness of message-based rehabilitation on cardiometabolic risk factors for PAD patients who have received surgical revascularization. The transtheorectical model (TTM) [11] will be used as a framework for conceptualizing the process of behavior change. This model is well-suited to this messaging-based intervention as it allows understanding of participants' processes and dynamics of behavioral changes.

2. Aim This single-blinded randomized controlled trial aimed to evaluate the effectiveness of the message-based rehabilitation on fasting low density lipoprotein (LDL) level, Ankle-Brachial Index (ABI), healthy lifestyle behaviours, quality of life and smoking status for PAD patients who have received revascularization.

3. Research hypothesis The research hypothesis is that the message-based rehabilitation program improve the LDL, ABI and the cardiometabolic risk factors of peripheral artery disease (PAD) patients who have received revascularization.

4. Methodology 4.1 Study design This pilot randomised controlled trial aimed at examining the effectiveness of message-based lifestyle intervention. Peripheral artery disease patients who have received revascularization in the past 6 months, are randomized into 2 groups. The total sample size will be 160. Both intervention and control groups will receive face-to-face lifestyle adherence counseling and booklets at baseline. The intervention group will receive 4 mobile phone messages per week for 24 weeks. The messages are motivational advice to support lifestyle behavioral modification in various stages of behavioral changes. All participants will be follow up at 6-week and 6-month in Surgical Out Patient Department. Participants' ABI, lifestyle behaviors and quality of life will be assessed at baseline, 6- week and 6-month follow-up. Participants' fasting low density lipoprotein (LDL) level at baseline and at 6-month follow up will be retrieved from Computer Management System with approval of Dr. Leung Siu-kee, Chief Of Service Department of Surgery Tuen Mun Hospital. At least ten participants from intervention group will be purposively selected for individual face-to-face semi-structured interview to evaluate the mobile phone-based rehabilitation program at 6-month follow-up.

4.2 Study outcomes

Primary outcomes:

- Fasting blood low density lipoprotein (LDL) level

Secondary outcome:

* Smoking status
* Readiness for behavioural changes
* Health related Quality of life
* Self-reported walking physical exercise (session per week)
* Self-reported serving fruits and vegetables consumed per day
* BMI
* Fasting glucose level
* HDL level
* Total cholesterol level
* ABI

4.3 Study setting The study will be conducted in the Department of Surgery in Tuen Mun Hospital

4.4 Sampling method Probability sampling (simple random sampling) will be adopted for this study. Simple individual randomization method by sequentially numbered, opaque sealed envelopes (SNOSE) will be used to ensure the PI and participants will be concealed from the allocation sequence. The trained research assistant will prepare 160 identical, opaque, sealed, A5-sized envelops, with a unique 3-digit serial number on the cover of each envelope as an identifier. Half of them will each contain a card indicating "intervention" and the other half, " control". After consent, the trained research assistant will open an envelope according to the sequence of the serial number and assign participant to either "intervention" or "control" group. The envelop must be opened according to the serial number. All others will not know the group allocation before the envelope is opened. Frequent checks (at least weekly) of these numbers will be done to ensure no deviation.

4.5 Sample size Sample size will be determined according to power (1-β), type 1 error (α), and effect size. The mean effect size of lifestyle intervention from a previous study is 0.4, which is a medium effect size according to Cohen 1998 [12]. Thus, an effect size of 0.4 was used in the calculations. To achieve the conventional level of 80% power and α= 5%, the sample size will be 128. The attrition rate in previous studies ranged from 16%-20%. A total of 160 participants will ultimately be required; 80 participants will be randomized to either intervention or control group.

4.6 Study intervention The message-based lifestyle intervention consists of three parts. Both the intervention and control groups will receive Parts I and II. Only the intervention group will receive Part III, which is the mobile phone messaging.

Part I: Conduct an individualized healthy lifestyle education The first part is face-to-face individual health education with supportive brief counselling. It consists of the identification of lifestyle risk factors and modification strategies for secondary prevention of PAD. This counselling service will be provided by Site Supervisor, Mr. Ng Hoi Wa. A measurable and realistic lifestyle modification plan will be established together with the client and the site supervisor.

Part II: Develop a healthy lifestyle booklet The second part is a reinforcement tool for face-to-face education. The research team will develop a booklet includes misconceptions, maladaptive beliefs, facilitators and barriers of healthy lifestyle modification.

Part III: Perform mobile phone-based messaging The trained research assistant will deliver the messages to the participants of the intervention group for 24 weeks throughout the study. The messages will act as a reinforcement to increase self-awareness about health-promoting behaviour and develop the desire for competence in achieving a healthy lifestyle.

5. Data collection The quantitative data will be collected by using questionnaires. The trained research assistant will explain the nature and purpose of the research to the potential participants in interview room in Department of Surgery. The eligible participants are requested to sign the informed-consent forms and reminded that their participation is voluntary. The participants are also requested to fill in two questionnaires, Patient Activation Measure [13] & Short Form 12 version 2 (SF12v2) [14], at the baseline, 6-week and 6-month follow-up. The participants' blood result of fasting low density lipoprotein (LDL) level will be retrieved from computer management system in Department of Surgery. Face-to-face individual semi-structured interviews will be conducted to collect qualitative data.

6. Data analysis Quantitative data will be analysed using International Business Machines Corporation(IBM) Statistics is leading statistical software (SPSS) version 22.0 [15]. The descriptive measures of all participants will be summarised by percentage, mean, and 95% confidence interval (CI), as well as compared for between-group differences. The t-test will be conduct to compare the differences in continuous variables between the intervention and control groups.

The qualitative data will be audio-recorded and analysed by thematic analysis. Seven open-ended questions will be used in the semi-structured interviews.

1. How do you feel about the mobile phone text message-based rehabilitation?
2. What factors encouraged you to participate in Peripheral Artery Disease Rehabilitation program?
3. What factors discouraged you from participate in Peripheral Artery Disease Rehabilitation program?
4. How did the mobile phone text message-based rehabilitation facilitate your participation in lifestyle modification?
5. How easy did you find following the lifestyle advice from the mobile phone text message?
6. How difficult did you find following the lifestyle advice from mobile phone text message?
7. Any suggestions on how to improve and promote the rehabilitation for patients with peripheral artery disease?

ELIGIBILITY:
Inclusion Criteria:

Aged above 50 Clinical diagnosis of peripheral artery disease Received revascularization in the past 6 months. Must be able to receive and read Chinese messages from their own mobile phones Must be able to come back for a 6-week and 6-month follow-up for lifestyle counselling and blood sample taking.

Exclusion Criteria:

Refuse to provide an informed-consent form. Clinical diagnosis of lack of capacity to provide informed consent.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of Fasting blood low density lipoprotein (LDL) level | Change from the baseline and 6-month follow-up.
  Fasting blood low density lipoprotein (LDL) level

SECONDARY OUTCOMES:
Change of Smoking status | Change from baseline, 6- week and 6-month follow-up
  self-reported 7-day point prevalence abstinence and validated by exhaled carbon monoxide monitor (<4 ppm)
Change of Readiness for behavioural changes | Change from baseline, 6- week and 6-month follow-up
  Measured by Patient Activation Measure
Change of Health related Quality of life | Change from baseline, 6- week and 6-month follow-up
  Measured by SF12v2
Change of BMI | Change from baseline, 6- week and 6-month follow-up
  Body Mas Index
Change of ABI | Change from baseline, 6- week and 6-month follow-up
  Ankle-Brachial Index
Change of Fasting glucose level | Change from baseline and 6-month follow-up
  Fasting glucose level
Change of HDL level | Change from baseline and 6-month follow-up
  HDL level
Change of Total cholesterol level | Change from baseline and 6-month follow-up
  Total cholesterol level

CONTACTS AND LOCATIONS:
Overall Officials: Hau Kim CHOY, MSc, Principal Investigator — Caritas Institute of Higher Education
Locations (2):
- Choy Hau Kim, Hong Kong, China
- Choy Hau Kim, Hong Kong, HK, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] European Stroke Organisation; Tendera M, Aboyans V, Bartelink ML, Baumgartner I, Clement D, Collet JP, Cremonesi A, De Carlo M, Erbel R, Fowkes FG, Heras M, Kownator S, Minar E, Ostergren J, Poldermans D, Riambau V, Roffi M, Rother J, Sievert H, van Sambeek M, Zeller T; ESC Committee for Practice Guidelines. ESC Guidelines on the diagnosis and treatment of peripheral artery diseases: Document covering atherosclerotic disease of extracranial carotid and vertebral, mesenteric, renal, upper and lower extremity arteries: the Task Force on the Diagnosis and Treatment of Peripheral Artery Diseases of the European Society of Cardiology (ESC). Eur Heart J. 2011 Nov;32(22):2851-906. doi: 10.1093/eurheartj/ehr211. Epub 2011 Aug 26. No abstract available. PMID 21873417
- [Result] Rantner B, Kollerits B, Pohlhammer J, Stadler M, Lamina C, Peric S, Klein-Weigel P, Muhlthaler H, Fraedrich G, Kronenberg F. The fate of patients with intermittent claudication in the 21st century revisited - results from the CAVASIC Study. Sci Rep. 2017 Apr 3;8:45833. doi: 10.1038/srep45833. PMID 28367968
- [Result] Hankey GJ, Norman PE, Eikelboom JW. Medical treatment of peripheral arterial disease. JAMA. 2006 Feb 1;295(5):547-53. doi: 10.1001/jama.295.5.547. PMID 16449620
- [Result] Khan S, Cleanthis M, Smout J, Flather M, Stansby G. Life-style modification in peripheral arterial disease. Eur J Vasc Endovasc Surg. 2005 Jan;29(1):2-9. doi: 10.1016/j.ejvs.2004.09.020. PMID 15570264
- [Result] Gerhard-Herman MD, Gornik HL, Barrett C, Barshes NR, Corriere MA, Drachman DE, Fleisher LA, Fowkes FG, Hamburg NM, Kinlay S, Lookstein R, Misra S, Mureebe L, Olin JW, Patel RA, Regensteiner JG, Schanzer A, Shishehbor MH, Stewart KJ, Treat-Jacobson D, Walsh ME. 2016 AHA/ACC Guideline on the Management of Patients With Lower Extremity Peripheral Artery Disease: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2017 Mar 21;135(12):e686-e725. doi: 10.1161/CIR.0000000000000470. Epub 2016 Nov 13. PMID 27840332
- [Result] Goel K, Lennon RJ, Tilbury RT, Squires RW, Thomas RJ. Impact of cardiac rehabilitation on mortality and cardiovascular events after percutaneous coronary intervention in the community. Circulation. 2011 May 31;123(21):2344-52. doi: 10.1161/CIRCULATIONAHA.110.983536. Epub 2011 May 16. PMID 21576654
- [Result] Dunlay SM, Witt BJ, Allison TG, Hayes SN, Weston SA, Koepsell E, Roger VL. Barriers to participation in cardiac rehabilitation. Am Heart J. 2009 Nov;158(5):852-9. doi: 10.1016/j.ahj.2009.08.010. Epub 2009 Sep 29. PMID 19853708
- [Result] Chow CK, Redfern J, Hillis GS, Thakkar J, Santo K, Hackett ML, Jan S, Graves N, de Keizer L, Barry T, Bompoint S, Stepien S, Whittaker R, Rodgers A, Thiagalingam A. Effect of Lifestyle-Focused Text Messaging on Risk Factor Modification in Patients With Coronary Heart Disease: A Randomized Clinical Trial. JAMA. 2015 Sep 22-29;314(12):1255-63. doi: 10.1001/jama.2015.10945. PMID 26393848
- [Result] Pfaeffli Dale L, Whittaker R, Jiang Y, Stewart R, Rolleston A, Maddison R. Text Message and Internet Support for Coronary Heart Disease Self-Management: Results From the Text4Heart Randomized Controlled Trial. J Med Internet Res. 2015 Oct 21;17(10):e237. doi: 10.2196/jmir.4944. PMID 26490012
- [Result] Hong Kong Census and Statistics Department: Information Technology usage 2016. Retrieved from https://www.censtatd.gov.hk/hkstat/sub/gender/itu/index.jsp.
- [Result] Prochaska JO, Velicer WF. The transtheoretical model of health behavior change. Am J Health Promot. 1997 Sep-Oct;12(1):38-48. doi: 10.4278/0890-1171-12.1.38. PMID 10170434
- [Result] Cohen J. Statistical power analyses for the social sciences. Hillsdale, NJ, Lawrence Erlbauni Associates. 1988.
- [Result] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Result] Wagner III WE. Using IBM® SPSS® statistics for research methods and social science statistics. Sage Publications; 2014 Mar 20.
- [Result] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939